CLINICAL TRIAL: NCT00287157
Title: A Double-Blind, Randomized, Two-Way Crossover, Comparative Study to Evaluate the Clinical Efficacy and Safety of Novel Sublingual Tizanidine HCl Versus Placebo in Children With Chronic Traumatic Brain Injury
Brief Title: Pilot, Proof-of-Concept Study of Sublingual Tizanidine in Children With Chronic Traumatic Brain Injury (TBI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva GTC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol C2/5/TZ-TBI-01
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Actigraphy; Spasticity, Cognition and Functioning
MeSH Terms: conditions — Brain Injuries, Traumatic; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Sublingual Tizanidine HCl

SUMMARY:
Nightly administration of a unique, sublingual (under the tongue) formulation of tizanidine, a known anti-spasticity medication, has been shown in a previous study to improve sleep and next-day functioning in CP (cerebral palsy) patients. It is hypothesized that this improvement in sleep efficiency (i.e.,fewer wake episodes, longer time asleep, etc.) with resulting improvement in quality-of-life (i.e.,improvements in next-day functioning, cognition and movement) may also be seen in a similar patient population, i.e., children with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Sublingual tizanidine, a novel test formulation of the known effective antispasticity agent, has been shown to have a unique pharmacokinetic profile [(i.e., nearly twice the bioavailability/AUC), but with little or no increase in peak plasma levels (Cmax), as compared to oral tizanidine (Zanaflex)]. When administered nightly to CP (Cerebral Palsy) patients to more effectively reduce the muscle spasms that disrupt sleep, it was shown to improve sleep efficiency, decrease sleep fragmentation and improve the sleep cycle. This improvement in night-time sleep was translated into a potential improvement in next-day functioning (improvement in next-day measures of spasticity and movement).

It is hypothesized that a similar type of improvement in sleep with consequent positive impact on next day improvement in spasticity, cognition and function, may also be manifest in a similar patient population, children with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Males/Females 8-18 years of age with documented history of TBI
* Documented Loss of Consciousness(LOC) for more than 24 H, or initial GCS (Glasgow Coma Score) lower than 8
* Current Spasticity that interferes with task performance
* Patient is able to cooperate and understand general explanations

Exclusion Criteria:

* History of allergy to tizanidine or any inactive component (including lactose intolerance)
* Use of other hypnotic medication within 3 days of baseline visit and during the study
* Botox therapy within 6 weeks of baseline, or use of Baclofen pump during the trial
* Use of CYP1A2 inhibitors (ex. ciprofloxacin or fluvoxamine) for the duration of the study
* Female patients on oral contraceptives
* Significant abnormalities in clinical screening laboratory parameters (ALT, AST, Bilirubin>2 x uln; Creatinine>2 mg/dl;WBC <2300/mm3, platelets<80,000/mm3)
* Taking of other medications that may adversely interfere with the actions of the study medication or outcome variables within 2 weeks of 5 half-lives of the baseline visit

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Improvement in Spasticity, Cognition and Daily Function | 4 weeks

SECONDARY OUTCOMES:
Improvement in nighttime actigraphy sleep parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ido Yatsiv, MD, Principal Investigator — Hadassah Medical Center, Ein Kerem, Jerusalem
Locations (1):
- Alyn Hospital Pediatric and Adolescent Rehabilitation Center, Jerusalem, Israel